CLINICAL TRIAL: NCT03645369
Title: The Effectiveness of Mechano-Analgesia and Cold Application
Brief Title: Effectiveness of Mechano-Analgesia and Cold Application on Ecchymosis, Pain and Satisfaction at Subcutaneous Heparin Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Demet İnangil, PhD, Principal Investigator, Istanbul Saglik Bilimleri University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 108400987-67
Record Dates: First submitted 2018-08-09; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Injection Site Reaction; Injection Site Bruising
Keywords: subcutaneous heparin; injection pain; ecchymosis
MeSH Terms: conditions — Injection Site Reaction; Ecchymosis

STUDY DESIGN:
Who Masked: Participant
Masking Description: This study was conducted on receiving treatment patients in the Orthopedics and Traumatology wards of a university hospital.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mechano-Analgesia (Experimental): The first SC heparin injections were applied from the right abdominal region using ShotBlocker®.
  Interventions: Device: ShotBlocker
- Cold Application (Experimental): The second SC heparin injections were applied from the left abdominal region with an ice pack
  Interventions: Device: Ice pack
- Control (No Intervention): The second SC heparin injections were applied from the lower abdominal region without any additional application

INTERVENTIONS:
Device: ShotBlocker — ShotBlocker is a drug-free tool with no side effects and does not require preparation. It is a flexible, plastic, C-shaped device with a number of short (2 mm) blunt contact points on its back.
  Arms: Mechano-Analgesia
Device: Ice pack — Ice pack containing gel
  Arms: Cold Application

SUMMARY:
Fifty-five patients received three subcutaneous heparin injections (165 injections) by the same investigator using additional techniques such as mechano-analgesia and cold application, and without any additional techniques.

DETAILED DESCRIPTION:
The abdomen was divided into four quarters. The first, second, and third SC heparin injections were applied from the right abdominal region using ShotBlocker®, left abdominal region with an ice pack, and lower abdominal region without any additional application, respectively. All the injection sites were circled using a skin marking pen (r = 5 cm).

All the injections were administered following a standard procedure. Pain and satisfaction were assessed immediately after the injection by using the VAS score. Ecchymosis was assessed with an ecchymosis measurement tool at 48 and 60 hours after the injection (Figure 3).

ELIGIBILITY:
Inclusion Criteria:

* Must be older than 18 years
* Open to communication
* No complications during the operation
* Normal body mass index (BMI; reference range, 18.5-29.9 kg/m2) (d) and
* Platelet count (150.000-300.000)
* Give consent to participate in the study

Exclusion Criteria:

* Oral and parenteral anticoagulant treatment for at least 5 days
* Infection, scar tissue or incision, and parenteral treatment in their abdominal area
* Hematological and allergic disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2015-03-15 (Actual); Study Completion 2015-12-25 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Measure via VAS | Immediately after injection
  The VAS was used to measure pain intensity. The VAS was composed of a 10-cm long line, which had subjective descriptive expressions on both sides (0 cm: no pain and 10 cm: unbearable pain). The individual was asked to make a sign on the line indicating the degree of the pain. The numerical values were recorded by the researcher.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Celik N, Khorshid L. The Use of ShotBlocker for Reducing the Pain and Anxiety Associated With Intramuscular Injection: A Randomized, Placebo Controlled Study. Holist Nurs Pract. 2015 Sep-Oct;29(5):261-71. doi: 10.1097/HNP.0000000000000105. PMID 26263287